CLINICAL TRIAL: NCT06090786
Title: A Multicentric, Prospective Study Addressing the Kinetics and Impact on Survival of Measurable Residual Disease in Acute Myeloid Leukemia Patients Receiving Azacitidine and Venetoclax
Brief Title: Kinetics and Impact on Survival of MRD in AML Patients Receiving Azacitidine and Venetoclax
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AML2723
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: AML, Adult; Minimal Residual Disease
Keywords: Venetoclax; Azacitidine; AML; Minimal rsidual disease
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRD evaluation (Other): Evaluation of MRD at pre-defined timepoints in AML patients treated with Azacitidine and Venetoclax
  Interventions: Diagnostic Test: MRD assessment

INTERVENTIONS:
Diagnostic Test: MRD assessment — Bone marrow withdrawal for MRD quantification

SUMMARY:
The goal of this no-profit, multicenter, biological, non-pharmacologic study is to evaluate minimal residual disease (MRD) in patients treated with Azacitidine and Venetoclax according to clinical practice.

The main questions it aims to answer are:

1. kinetics of disease response on treatment with Azacitidine and Venetoclax through the evaluation of MRD with both cytofluorimetric and molecular techniques
2. impact of MRD on survival outcomes. To this end, bone marrow samples will be collected at pre-defined time-points during treatment and MRD will be assessed.

DETAILED DESCRIPTION:
This is a multicentric biological study at evaluating MRD kinetics during treatment with Azacitidine and Venetoclax as well as the impact of MRD on survival outcomes.

Newly diagnosed, previously untreated, patients with AML, including de novo, secondary and therapy-related, receiving front-line therapy with Azacitidine and Venetoclax according to clinical practice will be included.

Response assessment will be performed on BM aspirate according to ELN2022 response criteria. MRD evaluation will be performed on BM at pre-defined time-points during treatment. MRD assessment will be performed centrally in order to harmonize response evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 18 years of age
* Subject has diagnosis of AML according to WHO 2016
* Subject has newly diagnosed, previously untreated, AML, including de novo, secondary and therapy-related (cytoreduction with hydroxyurea is admitted prior treatment start)
* Subject is planned to receive front-line therapy with Azacitidine and Venetoclax
* Subject is ineligible for intensive induction chemotherapy according to investigator assessment according to clinical practice
* Subject must have assessable MRD by flow cytometry at screening BM evaluation
* Signed written informed consent according to ICH/EU/GCP and national local laws

Exclusion Criteria:

* Diagnosis of BCR::ABL1-positive AML
* Diagnosis of APL
* AML with CNS involvement.
* AML with extra-medullary localizations
* Patients' unwillingness or inability to comply with the protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Rate of MRD-negative patients within cycle 4 | 4 months
  Number of patients without minimal residual disease within cycle 4 on the total of subjects receiving at least one dose of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Curti, Principal Investigator — Division of Hematology IRCCS Azienda Ospedaliero-Universitaria di Bologna

IPD SHARING:
Plan to Share IPD: No